CLINICAL TRIAL: NCT05520047
Title: Assessment and Prognostic Factors of Long-term Quality of Life of Patients Hospitalized With Severe COVID-19 and Their Relatives
Brief Title: Long-term Quality of Life and Prognostic Factors in Severe COVID-19 Patients and Their Relatives
Acronym: QUALICOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02Obs-CHRMT
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; Quality of Life; Posttraumatic Stress Disorder; Cognitive Impairment; Social Behavior
MeSH Terms: conditions — COVID-19; Stress Disorders, Post-Traumatic; Cognitive Dysfunction; Social Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID19-severe Patient: modified Medical Research Council dyspnea scale (mMRC), European Quality of Life 5 Dimensions and 5 Lines (EQ-5D-5L), the impact of event scale-revised (IES-R), The Hospital Anxiety and Depression Scale (HADS), the Montreal Cognitive Assessment (MoCA)- BLIND, Lawton instrumental activities of daily living (IADL) and Return to work scales
  Interventions: Behavioral: COVID19-severe Patient
- family of COVID19-severe Patient: impact of event scale-revised (IES-R), The Hospital Anxiety and Depression Scale (HADS) scales
  Interventions: Behavioral: family of COVID19-severe Patient

INTERVENTIONS:
Behavioral: COVID19-severe Patient — Behavioral and social test assessment
  Groups: COVID19-severe Patient
Behavioral: family of COVID19-severe Patient — Behavioral and social test assessment
  Groups: family of COVID19-severe Patient

SUMMARY:
This is a prospective cohort study with multicenter retrospective data collection (CHR Metz-Thionville, Hôpital Mercy and Hôpital Bel Air).

Patients hospitalized for COVID-19 in a critical care unit between March 2020 and March 2022 will be contacted by telephone 24 months after their hospitalization by a doctor or intern from the intensive care unit. If the patient agrees to participate, he or she will then complete the study questionnaire items. Data concerning their hospital management between their hospitalization for COVID-19 and the 24-month call will then be extracted from their medical records.

DETAILED DESCRIPTION:
The first wave of the global SARSCoV2 pandemic in March and April 2020 hit many regions of the world hard, including our Grand Est region, which had to reorganize its healthcare system in an emergency and in an unprecedented manner. The morbidity and mortality linked to this 1st wave is already very high, with mortality in intensive care units reaching 40% in the most affected regions.

Mortality, particularly in the short term, has long been the cornerstone of critical care evaluation. The development of resuscitation techniques in recent years has led to a substantial improvement in the survival of more and more patients, but also older and more polypathological patients. However, this hard criterion of mortality seems nowadays a little obsolete, making it prefer on the one hand the evaluation of the mortality in the longer term, but also and especially the evaluation of the quality of this survival. The interest has therefore shifted in recent years towards the long-term evaluation of criteria more focused on the patient but also on the family. Current data in pathologies such as Acute respiratory distress syndrome (ARDS) or severe sepsis concur to show that these are invariably associated with an alteration in quality of life, in all the domains of its original definition by the World Health Organization (WHO), and are at the origin of a "post-resuscitation syndrome".

COVID19 is marked in 5 to 10% of cases by a severe septic picture, with multivisceral dysfunction, and pulmonary involvement in the foreground. The existence of so-called "long COVID" clinical pictures already described in the literature and the media, and especially the obvious arrival of a second wave and perhaps others, make it necessary to study the long-term prognosis of this emerging infection.

The aim of this work is to quantify in a multimodal way the long-term quality of life of patients surviving a severe form of COVID19 and their families and to try to identify elements related to the patient, the COVID19, or the management, which predict this quality of survival. The theme concerned is on the one hand epidemiological and risk assessment for the populations, and on the other hand preventive and curative of late sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Having stayed in a critical care unit (resuscitation, continuous monitoring, intensive care) at the Regional Hosiptal Center (CHR) Metz-Thionville for COVID-19 between March 2020 and March 2022
* Having given their oral consent to participate (telephone contact), or not having objected during their lifetime to the use of their hospital data for epidemiological research (deceased patients)
* The trusted person or closest family member will also be invited to participate.
* The patients included will be those who were hospitalized in conventional critical care services, but also in functional units of so-called "ephemeral" critical care, armed in emergency in the context of a massive influx of victims (Cardiological Intensive Care, Post-Interventional Monitoring Room in the operating room, Dialysis Center).

Exclusion Criteria:

* Patient under guardianship or deprivation of liberty
* Cognitive disorders or lack of French language skills preventing response to evaluation questionnaires

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 severe patients
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Quality of life at 2 years in patients hospitalized in the Critical Care Unit for COVID-19 | 2 years after hospitalization for severe COVID-19
  The quality of life score at 2 years is assessed using the European Quality of Life 5 Dimensions and 5 Lines (EQ-5D-5L) questionnaire: it is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
  5 dimensions of the EQ-5D-5L scale. The dimensions assessed are: mobility, autonomy, impact on daily activities, pain and discomfort, and anxiety and depression.
  Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

SECONDARY OUTCOMES:
Dyspnea in patients hospitalized in the Critical Care Unit for COVID-19 using Modified Medical Research Council (mMRC) Dyspnea Scale | 2 years after hospitalization for severe COVID-19
  Modified Medical Research Council (mMRC) Dyspnea Scale : is recommended for conducting assessments of dyspnea and disability and functions as an indicator of exacerbation. The mMRC questionnaire is a 5-point scale and asks patients to rate dyspnea from 0 (absent) to 4 (dyspnea when dressing/undressing)
Mortality in patients hospitalized in the Critical Care Unit for COVID-19 | 2 years after hospitalization for severe COVID-19
  Vital status collected in hospital data or in public data from the French Institute of Statistics and Economic studies (INSEE)
Satisfaction/quality of life in patients hospitalized in the Critical Care Unit for COVID-19 | 2 years after hospitalization for severe COVID-19
  5 dimensions of the EQ-5D-5L scale. The dimensions assessed are: mobility, autonomy, impact on daily activities, pain and discomfort, and anxiety and depression.
  Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Posttraumatic stress in patients hospitalized in the Critical Care Unit for COVID-19 | 2 years after hospitalization for severe COVID-19
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score.
  Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case.
Cognitive impact in patients hospitalized in the Critical Care Unit for COVID-19 using The Montreal Cognitive Assessment (MoCA)- BLIND questionnaire | 2 years after hospitalization for severe COVID-19
  The Montreal Cognitive Assessment (MoCA)- BLIND is an adapted version of the original MoCA, a rapid screening instrument for mild cognitive dysfunction. The MoCA-BLIND assesses different cognitive domains: attention and concentration, memory, language, conceptual thinking, calculations, and orientation. It contains the same items as the original MoCA except those requiring visual abilities have been removed. Time to administer the MoCA- BLIND is approximately 5-10 minutes. The total possible score is 22 points; a score of 18 or above is considered normal. This cutoff score is suggestive as it has not been validated thus far.
Social and professional impact in patients hospitalized in the Critical Care Unit for COVID-19 using Lawton INSTRUMENTAL ACTIVITIES OF DAILY LIVING SCALE (IADL) | 2 years after hospitalization for severe COVID-19
  Lawton INSTRUMENTAL ACTIVITIES OF DAILY LIVING SCALE (IADL) questionnaire. The Lawton IADL scale takes 10 to 15 minutes to administer and contains eight items, with a summary score from 0 (low function) to 8 (high function). The scale can be administered with a written questionnaire or by interview. The patient or a knowledgeable family member or caregiver may provide answers.
Post-traumatic stress in the family of patients hospitalized in the Critical Care Unit for COVID-19 using the impact of event scale-revised (IES-R) questionnaire | 2 years after hospitalization for severe COVID-19
  impact of event scale-revised (IES-R) questionnaire assesses self-reported PTSD symptomatology experienced in the past 7 days, and consists of 22 items measured on a five point Likert scale (0-4, with labels of 'Not at all' to 'Extremely').
Post-traumatic stress in the family of patients hospitalized in the Critical Care Unit for COVID-19 using Hospital Anxiety and Depression Scale (HADS) questionnaire | 2 years after hospitalization for severe COVID-19
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score.
  Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case.

CONTACTS AND LOCATIONS:
Overall Officials: Damien BARRAUD, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No